CLINICAL TRIAL: NCT02965742
Title: Clinical Evaluation Of An X-Ray Bone Densitometer: Use Of DXA Technology For Precise Assessment Of Body Composition In Humans
Brief Title: Clinical Evaluation Of An X-Ray Bone Densitometer:Use Of DXA Technology For Precise Assessment Of Human Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diagnostic Medical Systems (Industry)
Collaborators: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00596-43
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Osteodensitometry
Keywords: DXA; DMS; DMS Imaging; STRATOS; Horizon A; QDR4500A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The study population: first 25 patients (Experimental): The study population consists of patients referred to the Nuclear Medicine and Medical Biophysics Department of the Montpellier University Hospital for the performance of an osteodensitometric examination.
  Intervention: Whole body and sub-regions exams using the "Stratos" Intervention: Whole body and sub-regions exams using the "Hologic QDR 4500A" Intervention: Whole body and sub-regions exams using the "Hologic HORIZON A"
  Interventions: Device: Stratos; Device: "Hologic QDR 4500A"; Device: "Hologic HORIZON A"
- The study population: last 25 patients (Experimental): The study population consists of sportsmen patients referred to the Nuclear Medicine and Medical Biophysics Department of the Montpellier University Hospital for the performance of an osteodensitometric examination.
  Intervention: Whole body and sub-regions exams using the "Stratos" Intervention: Whole body and sub-regions exams using the "Hologic QDR 4500A" Intervention: Whole body and sub-regions exams using the "Hologic HORIZON A"
  Interventions: Device: Stratos; Device: "Hologic QDR 4500A"; Device: "Hologic HORIZON A"

INTERVENTIONS:
Device: Stratos — A machine made by DMS group.
Device: "Hologic QDR 4500A" — A machine made by Hologic inc.
Device: "Hologic HORIZON A" — A machine made by Hologic inc.

SUMMARY:
The main objectives of this study are:

* to assess the concordance of body composition measures between two bone densitometry devices: the STRATOS by Diagnostic Medical Systems (DMS) and the Hologic QDR 4500 A by Hologic inc.
* to assess the concordance of body composition measures between two bone densitometry devices: the STRATOS by Diagnostic Medical Systems (DMS) and the Hologic HORIZON A by Hologic inc.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* the assessment of the consistency of body composition measurements at local level (arms, trunk, legs) between the Stratos and Hologic 4500 A,
* the assessment of the consistency of body composition measurements at local level (arms, trunk, legs) between the Stratos and Hologic HORIZON A,
* Monitoring the evolution of body composition in patients receiving at least two evaluations of DXA Hologic QDR 4500A on: patients treated for obesity or anorexia nervosa, sports people and other patient with prescription DXA and the assessment the consistency of body composition measurements in terms,
* Monitoring the evolution of body composition in patients receiving at least two evaluations of DXA Hologic HORIZON A on: patients treated for obesity or anorexia nervosa, sports people and other patient with prescription DXA and the assessment the consistency of body composition measurements in terms.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is referred by a doctor for the performance of an osteodensitometry examination or sportsmen coming through a protocol where the nuclear medicine department is the investigator center

Exclusion Criteria:

* The patient is pregnant or nursing
* The patient is unable to sign or refuse to sign the informed consent
* The patient has a coronary stent or metal sutures in the heart
* The patient has any type of metal objects in the body such as an artificial joint, a pin or a metal plate
* The patient has a pacemaker or defibrillator
* Patient weighing more than 200 kg or more than 2 meters high by 65 centimeters wide
* The patient is using an insulin pump or with insulin-necked
* The patient has undergone X-ray examination using a contrast medium such as barium in the previous seven days visit,
* Patient who underwent an examination using x rays in the 15 days preceding the visit
* Patient suffering from generalized edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Lin concordance coefficient | Day 0
  In order to get a first idea of the adequacy of the two techniques measurements of the two bone densitometers, a calculation of intraclass correlation coefficients will be done. To supplement this data, a correlation study between the two techniques will be performed. For this we will use the Bland-Altman technique and a study of LIN concordance correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Denis MARIANO-GOULART, Phd.Medecine, Principal Investigator — Nuclear department
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Undecided